CLINICAL TRIAL: NCT06767618
Title: Investigation of Upper Extremity Exercise Capacity, Hand Grip Strength and Daily Living Activities in Rheumatoid Arthritis Patients
Brief Title: Investigation of Upper Extremity Functions in Patients With Rheumatoid Arthritis
Status: Recruiting | Type: Observational
Sponsor: Kirsehir Ahi Evran Universitesi (Other)
Responsible Party: Principal Investigator, Başak KAVALCI KOL, Principal Investigator, Kirsehir Ahi Evran Universitesi
Other Study IDs: AhiEvranU525
Record Dates: First submitted 2025-01-06; First posted 2025-01-10 (Actual); Last update posted 2025-02-11 (Actual); Status verified 2025-02

CONDITIONS: Rheumatoid Arthritis
Keywords: exercise capacity; upper extremity; hand-grip strength
MeSH Terms: conditions — Arthritis, Rheumatoid

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Rheumatoid arthritis group: Rheumatoid arthritis patients in clinical remission between the ages of 18-75, who are followed up in the Kirsehir Ahi Evran University Physical Medicine and Rehabilitation Department outpatient clinic, will be included in the study.
- Control group: As a control group, healthy individuals between the ages of 18-75 years, who are similar to the patients in terms of age and gender, have no diagnosed disease, will be included in the study.

SUMMARY:
There are limited studies in the literature evaluating upper extremity functional exercise capacity, muscle functions and daily living activities in rheumatoid arthritis patients. In this context, the aim of this study was to investigate upper extremity exercise capacity, hand grip strength and daily living activities in rheumatoid arthritis patients.

DETAILED DESCRIPTION:
Rheumatoid arthritis is an inflammatory autoimmune chronic and systemic disease of unknown etiology. In addition to musculoskeletal involvement, lung involvement can also be observed in patients. Lung involvement and accompanying symptoms cause deterioration of physical function, quality of life and functional capacity. In rheumatoid arthritis, dyspnea can be observed during exertion due to disease progression, drug toxicity and respiratory/cardiovascular morbidities. In patients, decreased respiratory muscle strength, respiratory functions, carbon monoxide diffusion capacity and oxygen consumption also cause decreased physical functions. It has been reported that upper extremity exercise capacity and functional performance are reduced in patients with interstitial lung disease. It is known that peripheral muscle strength is an independent determinant of exercise capacity in interstitial lung disease. Rheumatoid cachexia, characterized by decreased muscle mass and increased fat mass, is observed in rheumatoid arthritis patients. Since the patients' accessory respiratory muscles are also affected, it can negatively affect their daily life activities, especially those that use the upper extremities.

ELIGIBILITY:
Inclusion Criteria:

Inclusion criteria for patients with rheumatoid arthritis

* Patients diagnosed with rheumatoid arthritis,
* Between the ages of 18-75 years,
* Patients who volunteer to participate in the study will be included in the study.

Inclusion criteria for the healthy control group

* Between the ages of 18-75 years,
* Volunteer to participate in the study will be included in the study.

Exclusion Criteria:

Exclusion criteria for patients with rheumatoid arthritis

* Those with serious cardiopulmonary, neurological, neuromuscular, orthopedic and other systemic diseases or other diseases affecting physical functions,
* Those who have participated in a planned exercise program in the last three months
* Those with cognitive impairment that will cause difficulty in understanding and following exercise test instructions
* Patients with contraindications for exercise testing or exercise training according to the American Sports Medicine Association will not be included in the study.

Exclusion criteria for the healthy control group

* Those with any diagnosed chronic or systemic disease,
* Those who smoke 10 packs x years or more,
* Those who have pneumonia or any acute infection,
* Healthy individuals with any psychiatric disorder will not be included in the study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Rheumatoid arthritis patients between the ages of 18-75 who are clinically in remission and are being followed up at the Kirsehir Ahi Evran University Physical Medicine and Rehabilitation Department polyclinic will be included in the study. As a control group, healthy individuals who are similar to the patients in terms of age and gender and do not have any disease will be included in the study.
Sampling Method: Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2025-01-25 (Actual); Primary Completion 2026-01-25 (Estimated); Study Completion 2027-01-25 (Estimated)

PRIMARY OUTCOMES:
Evaluation of Upper Extremity Exercise Capacity | First day and second day
  The six minute peg board and ring test will be used to assess upper extremity exercise capacity.
Glittre Activities of Daily Living | Second day
  The Glittre activities of Daily Living test will be used to evaluate the daily living activities of individuals.

SECONDARY OUTCOMES:
Hand-grip strength | First day
  Hand-grip strength will be assessed using a hand dynamometer.
Evaluation of upper extremity functional status | First day
  The Arm, Shoulder and Hand Disabilities Questionnaire (DASH) will be used to evaluate the upper extremity functional status of individuals. The DASH evaluates the functional status of the upper extremity subjectively according to the Likert scale. It consists of 3 sections. The questionnaire scores between 0 (no disability) and 100 (severe disability).
Evaluation of arm and shoulder muscle strength and endurance | Second day
  The Thirty-Second Push-Up Test will be used to evaluate arm and shoulder muscle strength and endurance.

CONTACTS AND LOCATIONS:
Overall Officials: Başak KAVALCI KOL, PhD, Principal Investigator — Kirsehir Ahi Evran Universitesi; Merve FIRAT, PhD, Study Chair — Kirsehir Ahi Evran Universitesi; Figen TUNCAY, Prof. Dr., Study Chair — Kirsehir Ahi Evran Universitesi
Locations (1):
- Kırşehir Ahi Evran University, Physical Therapy and Rehabilitation Center, Cardiopulmonary Unit, Kırşehir, Merkez, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Individual participant data will be stored in a locked cabinet.

REFERENCES:
- [Background] Palugan MJA, Assis ACB, Bessa EJC, Ferreira AS, Lopes AJ. Predictors of functional capacity as measured by the Glittre activities of daily living test in women with rheumatoid arthritis. Braz J Med Biol Res. 2021 Mar 15;54(5):e10040. doi: 10.1590/1414-431X202010040. eCollection 2021. PMID 33729387
- [Background] Higgins SC, Adams J, Hughes R. Measuring hand grip strength in rheumatoid arthritis. Rheumatol Int. 2018 May;38(5):707-714. doi: 10.1007/s00296-018-4024-2. Epub 2018 Apr 6. PMID 29626222